CLINICAL TRIAL: NCT04634383
Title: ICVP - A Phase I Clinical Trial to Determine the Feasibility of a Human Cortical Visual Prosthesis for People With Blindness
Brief Title: A Phase I Feasibility Study of an Intracortical Visual Prosthesis (ICVP) for People With Blindness
Acronym: ICVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Illinois Institute of Technology (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Rush University Medical Center (Other); The Chicago Lighthouse (Other); The University of Texas at Dallas (Other); University of Chicago (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ICVP0001; UH3NS095557 (NIH)
Record Dates: First submitted 2020-10-12; First posted 2020-11-18 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Ocular Injury; Optic Nerve Diseases; Photoreceptor Degeneration; Blindness,Acquired
Keywords: Blindness; Visual Prosthesis; Electrical Stimulation
MeSH Terms: conditions — Eye Injuries; Optic Nerve Diseases; Blindness

STUDY DESIGN:
Intervention Model Description: Eligible participants for the study will be persons with blindness who meet the listed inclusion criteria. Individuals having any of the listed exclusion criteria will not be eligible to participate in the study. Enrolled participants will receive electrical stimulation devices implanted in the cortical region of their brain that is involved in vision processing. A maximum of five participants will be implanted. Written Informed Consent will be obtained from all participants before they are enrolled in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- WFMA Cortical Visual Prosthesis Single-arm Study (Experimental): The WFMA is an electronic device that is implanted in the cortical vision processing regions of the brain to produce artificial vision.
  Interventions: Device: WFMA - wireless floating microelectrode array

INTERVENTIONS:
Device: WFMA - wireless floating microelectrode array — Wirelessly transmitted patterns of electrical stimulation will be delivered to the visual cortex of study participants to generate visual percepts.
  Other Names: ICVP System; ICVP; Intracortical Visual Prosthesis

SUMMARY:
The purpose of this study is to determine the feasibility of producing artificial vision in persons with blindness. Study participants will have wireless electrical stimulators implanted into the cortical vision processing areas of their brains. The ability of the participants to perceive artificial vision in response to electrical stimulation will be assessed.

DETAILED DESCRIPTION:
The objective of this study is to test the safety of the ICVP system and the feasibility of eliciting visual percepts in response to electrical stimulation in persons with blindness. The electrical stimulation is provided by wireless floating microelectrode arrays (WFMAs) that are part of the ICVP system. The WFMAs are implanted in the visual cortex. Five participants will take part in the study and each participant will have multiple WFMA devices implanted in their visual cortex on one side of the brain. After recovery from surgery, participants will begin a series of tests to assess the ability of electrical stimulation to induce visual percepts and how these percepts may provide some measure of artificial vision. Weekly participant testing will occur over a period of one to three years.

ELIGIBILITY:
Inclusion Criteria:

* No light perception or bare light perception, in each eye in accordance with relevant International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes, where the physician has no expectation of improvement through currently approved treatments.
* History of normal or near-normal vision, with or without refractive correction, during at least the first 10 years of life.
* Adjusted to blindness for at least one year.
* History of vision or blindness rehabilitation.
* Willing and able to meet the time demands of the study with transportation assistance.
* Willing to agree to audio and video recording, as specified in the pre-screening consent.
* Motivated by altruism, willingness to participate in pioneering science.
* Demonstrated support from spouse, family and/or friends.
* High or average cognitive and spatial functioning.
* Normal structural MRI.
* English as preferred language.
* Normal decision-making capacity.

Exclusion Criteria:

* Poor adjustment to blindness, or vision loss within the last year.
* Expectation of vision restoration to pre-blindness level through trial participation.
* History of alcohol or drug dependence.
* Evidence of prior immune response to an orthopedic implant which caused the implant to be explanted
* A disease prognosis of living less than five years.
* An implant which would prevent screening using MRI, or a pacemaker, or similar implant.
* A history of seizures.
* Current suicidal ideation.
* Poor decision-making capacity.
* Current diagnosis or history of severe mental illness.
* Women who are pregnant or plan on becoming pregnant in the duration of the trial.
* Hand Motion (HM) vision or better vision,
* No Light Perception (NLP) or Light Perception (LP) vision with present OptoKinetic Nystagmus (OKN)
* NLP vision with pupil constriction
* Patients with Islands of perceivable vision in Goldmann Visual Field or Confrontational visual Field will also be excluded from the study.
* Patients with Complete media opacity (complete cornea opacity, very dense cataract) that does not allow visualization of the posterior segment to determine the cause of blindness will be excluded from the study. Only patients with NLP and LP vision without OKN will be included in the study.
* Patients with NLP or LP vision since birth will also be excluded from the study, as they may not have fully developed higher visual pathways, including cortical connections

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
To test the safety of the WFMA-based cortical interface. | From two-weeks post-op to end of device use, up to 3 years.
  Safety is defined as the number of adverse events occurring over the study period due to surgical complications or use of the WFMA device.

SECONDARY OUTCOMES:
To test the efficacy of the WFMA-based cortical interface | From four-weeks post-op to end of device use, up to 3 years.
  Efficacy is defined as establishing a chronic intracortical interface for which the ability to elicit visual percepts in response to electrical stimulation can be demonstrated with stimulus intensities of 16 nanocoulombs per phase or less.

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Troyk, PhD, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Illinois Institue of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We may electively share de-identified study data with collaborators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Duration of the study
Access Criteria: Data required by study collaborators to perform analysis of safety and efficacy of the ICVP system.

REFERENCES:
- [Background] Bak M, Girvin JP, Hambrecht FT, Kufta CV, Loeb GE, Schmidt EM. Visual sensations produced by intracortical microstimulation of the human occipital cortex. Med Biol Eng Comput. 1990 May;28(3):257-9. doi: 10.1007/BF02442682. No abstract available. PMID 2377008
- [Background] Schmidt EM, Bak MJ, Hambrecht FT, Kufta CV, O'Rourke DK, Vallabhanath P. Feasibility of a visual prosthesis for the blind based on intracortical microstimulation of the visual cortex. Brain. 1996 Apr;119 ( Pt 2):507-22. doi: 10.1093/brain/119.2.507. PMID 8800945
- [Derived] Stephan K, Troyk PR, Dagnelie G, Cogan S, Barry MP, Grant P, Lane F, Szlyk JP, McNulty M, van Drongelen W, Pham TH, Stipp KL, Royster M, Towle VL. The Role of Scalp EEG Recordings During Cortical Visual Prosthesis Testing. Artif Organs. 2025 Sep;49(9):1417-1428. doi: 10.1111/aor.15023. Epub 2025 May 27. PMID 40421717